CLINICAL TRIAL: NCT04302636
Title: The Synergistic Effect of Hypoglycemic Index Diet on Refractory Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jijun Wang, professor of medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKM201919
Record Dates: First submitted 2020-03-08; First posted 2020-03-10 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Refractory Schizophrenia
Keywords: Schizophrenia; Low-glycemic Idex Diet
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The hypoglycemic index diet group (Experimental): Patients in the experimental group ate two portions of food each day.This diet will last for 12 weeks.
  1. Food provided by the canteen: one egg for breakfast;Lunch and dinner are 50g of rice with all the dishes.
  2. Dietary nutrition and supplementary food: according to the weight and height of the patient, the daily energy required was calculated, which was divided into six levels: 1400kcal, 1600kcal, 1800kcal, 2000kcal, 2200kcal and 2400kcal.The six corresponding nutritional auxiliary food powders are: 20g-30g-40g-50g-60g-70 g.The suspension was prepared in the proportion of 160ml warm water poured into 55 grams and given to the patient.
  Interventions: Dietary Supplement: Low glycemic index diet
- General diet group (No Intervention): The LGIT diet of the experimental group consisted of 55% fat, 30% protein and 15% carbohydrate, and the glycemic index of the food was limited to less than 50. The meal was prepared by a public nutritionist who evaluated the nutritional composition of the inpatients provided by the canteen and then added or subsumed the compound nutrition powder.

INTERVENTIONS:
Dietary Supplement: Low glycemic index diet — The LGIT diet of the experimental group consisted of 55% fat, 30% protein and 15% carbohydrate, and the glycemic index of the food was limited to less than 50. The meal was prepared by a public nutritionist who evaluated the nutritional composition of the inpatients provided by the canteen and then added or subsumed the compound nutrition powder.
  Arms: The hypoglycemic index diet group

SUMMARY:
This experiment was conducted to investigate the improvement of hypoglycemic index diet (LGIT) as a potential new intervention scheme for treatment-resistant schizophrenia, and to further explore the mechanism of efficacy.

DETAILED DESCRIPTION:
A low glycemic index diet (LGIT) is a modification of a ketogenic diet (KD) that includes low carbohydrate, medium protein, and high fat intake.It is a potential new intervention for refractory schizophrenia.The possible mechanism is that relatively low and stable blood sugar levels trigger the brain to start applying fat metabolism, helping to compensate for impaired GABA levels in the brain.KD can effectively treat refractory epilepsy, and its therapeutic effect on epilepsy is comparable to that of antiepileptic drugs, which have been written into the treatment guidelines as a good synergist and mood stabilizer in schizophrenia and various mental disorders.Therefore, it can be assumed that LGIT has a certain effect on the positive symptoms of schizophrenia as a synergistic agent.In this study, 80 patients with schizophrenia were randomly divided into two groups: LGIT diet and normal diet.The changes of PANSS and blood lipid before and after treatment were analyzed. Transcranial magnetic stimulation (TMS) was used to evaluate the gaba-mediated cortical excitability of patients to further explore the mechanism of efficacy.

Experimental design:

1)Experimental scheme:

1. Sample estimation and selection of cases: although not find LGIT to treat schizophrenia scale research for reference, but in an article published in 2018 KD the curative effect of treatment of refractory epilepsy in children and adherence of Meta analysis, Du Ailing from 1989 to 2018 were analyzed such as relevant information received 503 cases, termination of the experiments of the main causes of poor adherence to patients and family members, the loss rate of about 10%.Therefore, 80 cases meeting the inclusion criteria and exclusion criteria were included in this study, all of which were inpatients from huangpu district mental health center in Shanghai. The patients were divided into LGIT group (L) with 40 cases and normal diet group (N) with 40 cases by random number table method.
2. Inclusion criteria:

   * Meet the diagnostic criteria of schizophrenia in icd-10, and score ≥4 in any item of p1-7 in PANSS scale.

     ② Meet the diagnostic criteria for treatable schizophrenia: in the past 5 years to three drugs and the appropriate dose and course of antipsychotic drugs (three drugs at least two chemical structures are different) poor response; Adverse reactions of patients who cannot tolerate antipsychotic drugs; Even with adequate maintenance treatment or preventive treatment, the patient still relapses or deteriorates.

     ③ Age 18-65.
3. Exclusion criteria:

   * Patients with the following diseases: fatty acid transport or oxidation defects, ketone body synthesis or decomposition defects, mitochondrial diseases, serious liver diseases, pyruvate carboxylase defects, porphyria, carnitine deficiency, some immunodeficiency diseases, organic acid urine; ② Patients with bleeding tendency, severe hypertension and severe heart, liver, lung, kidney failure, severe epilepsy patients; ③ Serious history of alcohol and drug abuse, addiction; ④ Extremely excited restless patients;Patients using implantable electronic devices.
4. Withdrawal criteria:

   ① Complete the 12-week test process;

   ② LGIT patients in the experimental group and the normal diet control group continued to use the original drugs throughout the experiment. If the type or dose of antipsychotics changed due to the recurrence of the disease, they would withdraw from the experiment.

   ③ The patient can not tolerate the situation of diet treatment, autonomous request to withdraw.
5. Before treatment, at the end of the 4th week, the 8th week and the 12th week, venous blood was extracted from the elbow for four times, and the positive and negative symptom syndrome scale (PANSS), Hamilton anxiety scale (HAMA) and Hamilton depression scale (HAMD) were measured by two professional evalutors with blind evaluation.The neuropsychological state rating scale (RBANS) was used to assess changes in cognitive function before and after treatment.Transcranial magnetic stimulation (TMS) was used to assess changes in cortical excitability mediated by gaba-capable intermediate neurons in patients before and after treatment.
6. Efficacy evaluation criteria: according to obvious effect (PANSS score reduction rate >50%), effective (PANSS score reduction rate 25-50%), invalid (PANSS score reduction rate <25%).
7. the LGIT diet of the experimental group consisted of 55% fat, 30% protein and 15% carbohydrate, and the glycemic index of the food was limited to less than 50. The meal was prepared by a public nutritionist who evaluated the nutritional composition of the inpatients provided by the canteen and then added or subsumed the compound nutrition powder.

2)statistical treatment: SPSS21.0 statistical software package was used, measurement data were expressed as (x-±s), the mean level was 0.05, group t test was used for comparison before and after treatment, and correlation analysis was multiple stepwise regression analysis.

ELIGIBILITY:
1. Inclusion criteria:

   ①Meet the diagnostic criteria of schizophrenia in icd-10, and score ≥4 in any item of p1-7 in PANSS scale.

   ② Meet the diagnostic criteria for treatable schizophrenia: in the past 5 years to three drugs and the appropriate dose and course of antipsychotic drugs (three drugs at least two chemical structures are different) poor response; Adverse reactions of patients who cannot tolerate antipsychotic drugs; Even with adequate maintenance treatment or preventive treatment, the patient still relapses or deteriorates.
   * Age 18-65.
2. Exclusion criteria:

   * Patients with the following diseases: fatty acid transport or oxidation defects, ketone body synthesis or decomposition defects, mitochondrial diseases, serious liver diseases, pyruvate carboxylase defects, porphyria, carnitine deficiency, some immunodeficiency diseases, organic acid urine; ② Patients with bleeding tendency, severe hypertension and severe heart, liver, lung, kidney failure, severe epilepsy patients; ③ Serious history of alcohol and drug abuse, addiction; ④ Extremely excited restless patients;Patients using implantable electronic devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
PANSS score changes | 12 weeks
  Observe and record the patient's symptoms before dietary treatment and 4, 8, and 12 weeks of treatment. The PANSS score is used for evaluation. The lower the score, the better the effect is obtained.

SECONDARY OUTCOMES:
Changes in BMI | 12 weeks
  Measure the height of the patient, observe and record the weight change of the patient before the diet treatment and 12 weeks after the treatment, and calculate the BMI according to the formula "BMI (kg/m2)=weight (kg)/height (m)2". The closer the BMI is to the normal value, the better the effect obtained.

OTHER OUTCOMES:
Observe changes in total cholesterol | 12 weeks
  Before the diet treatment and after 12 weeks of treatment, test total cholesterol (mmol/L) and observe its changes.
Changes in RBANS score | 12 weeks
  Observe and record the changes in the patient's neuropsychological state before dietary treatment and after 12 weeks of treatment, and use RBANS for evaluation. The higher the score, the better the effect.
Observe changes in triglycerides | 12 weeks
  Before the diet treatment and after 12 weeks of treatment, test triglycerides (mmol/L) and observe its changes.
Observe changes in total serum protein | 12 weeks
  Before the diet treatment and after 12 weeks of treatment, test serum total protein (g/L), and observe its changes.
Observe changes in fasting blood glucose | 12 weeks
  Before the diet treatment and after 12 weeks of treatment, test fasting blood glucose (mmol/L), and observe its changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Huangpu District Mental Health Center, Shanghai, Shanghai Municipality, China